CLINICAL TRIAL: NCT02715336
Title: A Randomized Controlled Trial of Pre-retrieval Triggering Methods in in Vitro Fertilization Patients Classified as Low, Normal or High Responder
Brief Title: Efficacy and Safety of Medication Used to Stimulate Ovulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Create Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFC-01
Record Dates: First submitted 2016-03-05; First posted 2016-03-22 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: IVF Cycle; Ovarian Stimulation; Egg Retrieval; Pregnancy; Miscarriages; Ovarian Hyperstimulation
Keywords: In vitro fertilization; IVF; Assisted Reproductive Technologies; ART; OHSS; Ovarian hyperstimulation; dual triggering; GnRH
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Ovulation Induction; Leuprolide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Study group: High Responders (Experimental): 1000 units hCG
  Interventions: Drug: Ovulation induction with hCG and Lupron (GnRH agonist)
- Control group: High Responders (No Intervention): 1000 units hCG
- Study group: Normal Responders (Experimental): 5000 units hCG
  Interventions: Drug: Ovulation induction with hCG and Lupron (GnRH agonist)
- Control group: Normal Responders (No Intervention): 5000 units hCG
- Study group: Low Responders (Experimental): 10000 units hCG
  Interventions: Drug: Ovulation induction with hCG and Lupron (GnRH agonist)
- Control group: Low Responders (No Intervention): 10000 units hCG

INTERVENTIONS:
Drug: Ovulation induction with hCG and Lupron (GnRH agonist) — Patients treated for infertility are categorized as a low-, normal- or high responder according to their estimated ovarian response to hormonal stimulation. This classification dictates the hormonal stimulation regimen that they will receive. In contrast to hCG triggering, GnRHa triggering is characterized by simultaneous LH and FSH surges, similar to natural ovulation. A combination of GnRHa plus hCG for triggering creates simultaneous LH and FSH surges by the GnRHa, which resembles physiologic ovulation triggering, together with sustained LH-like activity from the hCG, stimulating the corpus luteum to excrete sufficient hormonal endometrial support.
  Arms: Study group: High Responders; Study group: Low Responders; Study group: Normal Responders

SUMMARY:
Individuals undergoing In Vitro Fertilization must undergo controlled ovarian hyperstimulation (COH) to produce enough quality eggs for fertility treatment. Ovarian follicular responsiveness to COH with gonadotropins is extremely variable between patients and even from cycle to cycle for the same patient. Achieving an ideal follicular response is critical to the success of assisted reproduction treatment (ART). Patients have been classified as 'poor', 'normal' or 'high' responders, which dictate the amount of gonadotropins that they receive. It is still important to develop treatments with high efficacy, lower multiple birth rates, and a lower complication rate for each of these groups. In an era of evidence-based medicine and with special emphasis on reducing IVF risks (mainly OHSS and pregnancies with multiples), it is very important to find optimal and safe ovulation induction and triggering regimens for each patient population.

The use of GnRH agonist (GnRHa) triggering among high responders in order to reduce or eliminate OHSS is an example of an important breakthrough in the clinical management of IVF patients. Although GnRHa triggering was shown to be as effective as human chorionic gonadotropin (hCG) at inducing oocyte maturation more than 20 years ago, its use to trigger ovulation was not possible until the introduction of GnRH antagonists for pituitary suppression.

Another prominent trend in ART in recent years has been the introduction of dual triggering, which involves a combination of GnRHa plus hCG for triggering. This regimen creates simultaneous lutenizing hormone (LH) and follicle stimulating hormone (FSH) surges by the GnRHa, which resembles physiologic ovulation triggering, together with sustained LH-like activity from the hCG, which stimulates the corpus luteum to excrete sufficient hormonal endometrial support. Since its introduction, dual triggering has been gaining popularity due to outstanding results in retrospective studies among both normal and high responders. Moreover, in spite of the encouraging retrospective reports, prospective randomized controlled trials (RCT) on dual triggering have not been reported to date. The aim of the current proposed study is to compare the efficacy of dual triggering and conventional triggering among the three IVF populations (high, normal and poor responders).

DETAILED DESCRIPTION:
Ovarian follicular responsiveness to controlled ovarian hyperstimulation (COH) with gonadotropins is extremely variable between patients and even from cycle to cycle for the same patient. Achieving an ideal follicular response is critical to the success of assisted reproduction treatment (ART). Since the early years of ART, patients have been classified as 'poor', 'normal' or 'high' responders. Although these terms are widely used in research and in daily clinical practice, their precise definitions are not fully agreed upon. Distinguishing them has been based on various measures of ovarian reserve. The first description of a poor responder occurred in 1983, and the first international consensus criteria for poor responders (the Bologna Criteria) was published in 2011. Poor responders, in general, exhibit an inadequate response to hormonal stimulation and diminished reproductive outcome. In contrast to poor responders, high responders are characterized by an exaggerated ovarian responsiveness, accompanied by a higher risk for ovarian hyperstimulation syndrome (OHSS). In most IVF clinics, "normal responders" comprise the majority of their patients. These patients are characterized by an adequate response to gonadotropins stimulation, a relatively low risk for OHSS, and a low cancellation rate. However, even with their relatively good prognosis, it is still important to develop treatments with high efficacy, lower multiple birth rates, and a lower complication rate. In addition, ovum donors are a unique population of patients with special characteristics and challenges. Egg donation has proven to be an effective treatment option for the treatment of various forms of infertility. However, ovum donors are a young population with a significant OHSS risk. Moreover, studies regarding this population provide an ideal opportunity to determine the effects of various triggering regimens on implantation (endometrial effect) from those attributable to the oocyte cohort alone (follicular effect). In an era of evidence-based medicine and with special emphasis on reducing IVF risks (mainly OHSS and pregnancies with multiples, it is very important to find optimal and safe ovulation induction and triggering regimens for each patient population. The use of GnRH agonist (GnRHa) triggering among high responders in order to reduce or eliminate OHSS is an example of an important breakthrough in the clinical management of IVF patients. Although GnRHa triggering was shown to be as effective as human chorionic gonadotropin (hCG) at inducing oocyte maturation more than 20 years ago, its use to trigger ovulation was not possible until the introduction of GnRH antagonists for pituitary suppression. In contrast to hCG triggering, GnRHa triggering is characterized by simultaneous LH and FSH surges, similar to natural ovulation. Early results with GnRHa triggering were disappointing, as reported in several RCT"s, where higher pregnancy loss rates and lower ongoing pregnancy rates were observed. Subsequently, outcomes were dramatically improved after the adoption of adjusted regimens to enhance luteal support. A pivotal study by Engmann et al (2008) included high responder patients during their first IVF cycle and patients with a history of high response in a previous cycle. The authors reported no cases of OHSS in those patients who underwent GnRHa triggering together with intensified estrogen and progesterone supplementation, while maintaining comparable reproductive outcome to those receiving HCG triggering. Moreover, increased safety of GnRHa triggering has been reported among ovum donors in several reports. Another well designed RCT, recruited patients with OHSS risk factors (PCOS as well as oligo/amenorrhea) and further differentiated them on the triggering day into "low" vs. "high" OHSS risk according to their actual ovarian response. These researchers emphasized the fact that pre-stimulation classification as a high responder does not optimally correlate with actual response to hormonal stimulation. Therefore, there is a need to distinguish between a) pre-stimulation assessment based on clinical, laboratory and ultrasonographic parameters (such as previous OHSS, anti-müllerian hormone (AMH) and antral follicle count (AFC), respectively) and b) the actual response evaluated by the number and size of recruited follicles and serum estradiol concentration. Another prominent trend in ART in recent years has been the introduction of dual triggering, which involves a combination of GnRHa plus hCG for triggering. This regimen creates simultaneous LH and FSH surges by the GnRHa, which resembles physiologic ovulation triggering, together with sustained LH-like activity from the hCG, which stimulates the corpus luteum to excrete sufficient hormonal endometrial support. Since its introduction, dual triggering has been gaining popularity due to outstanding results in retrospective studies among both normal and high responders. Griffin et al, 2012 reported that among high responders, their dual-trigger group (GnRHa plus 1,000 IU hCG) had a significantly higher live birth rate (52.9% vs. 30.9%), implantation rate (41.9% vs. 22.1%), and clinical pregnancy rate (58.8% vs. 36.8%) as compared to GnRHa alone, without a higher risk for OHSS. A large retrospective study, which included 376 normal responders patients with 378 completed cycles, resulted in a significantly higher implantation (29.6% vs. 18.4%), clinical pregnancy (50.7% vs. 40.1%), and live-birth (41.3% vs. 30.4%) rates with an hCG (6,500 IU) together with GnRH agonist, as compared to hCG alone. Additionally, dual triggering was found as efficient method to improve final oocyte maturation among patients with a high immature oocyte rate and in patients with a low number of oocytes retrieved per number of pre-ovulatory follicles. To the best of our knowledge, there are no reports on the effect of dual triggering on IVF outcome among poor responders or OHSS occurrence in ovum donors. Moreover, in spite of the encouraging retrospective reports, prospective RCTs on dual triggering have not been reported to date. The aim of the current proposed study is to compare the efficacy of dual triggering and conventional triggering among the three IVF populations (high, normal and poor responders), as well as ovum donors. The current proposal includes three different protocols, which will be implemented in four populations in separate simultaneous RCT's:

1. Dual triggering with 1000 units hCG vs. GnRH agonist alone in high responder IVF patients and in ovum donors.
2. Dual triggering vs. 5000 units hCG in normal responders
3. Dual triggering vs. 10000 units hCG in poor responders

ELIGIBILITY:
A) Dual triggering vs. GnRH agonist alone in high responders IVF patients

Inclusion Criteria - At least one of the following risk factors:

* AMH > 29 pmol/L
* AFC > 16
* PCOS diagnosed according to Rotterdam criteria: any two of the following three features: 1) oligo- or anovulation; 2) clinical and/or biochemical hyper-androgenemia; and 3) PCO-US with exclusion of other etiologies as mentioned in the National Institute of Child Health and Human Development (NICHD) criteria
* Previous OHSS
* Previous cycle cancellation due to OHSS risk
* Previous coasting
* Participants initially recruited to the normal responders study who exhibit excessive ovarian response markers on triggering day: high amount of middle-large follicles (> 13 follicles ≥ 11mm on triggering day). All previous inclusion criteria are assessed before initiation of the IVF cycle and ovarian stimulation, and all of them represent pre-stimulation risk factors for high ovarian response. The patient's actual response will be assessed on triggering day (after completion of ovarian stimulation). Final assignment of responder category followed by randomization will only be performed on the day of triggering
* informed consent obtained
* Must be 18 years or older
* Ability to speak and read English, or understand French, Mandarin, Cantonese, Arabic, or Filipino.

Exclusion criteria:

* Chronic disease
* Hypogonadotrophic hypogonadism
* Untreated uterine abnormalities
* E2>4000 pg/ml (>14,680 pmol/L) on trigger day. These very high risk patients will undergo GnRHa only trigger and will be excluded from the trial.

B) Dual triggering vs. 5000 units hCG in normal responders

Inclusion criteria:

* Age above 18 years and less than 40 years
* Do not fulfill criteria for poor responder or high responder

Exclusion criteria:

* Bologna criteria for poor responders exclusion: two of the following should need to be fulfilled:

  1. Age > 40 or other risk factor for decreased ovarian reserve (ex. ovarian surgery)
  2. Single abnormal test for ovarian reserve (AFC < 6 or AMH < 8 pmol/L)
  3. Previous poor response in previous cycle: cancellation or < 4 retrieved oocytes in response to daily 150 FSH units
* Criteria for high responders' exclusion

  1. AMH > 29 pmol/L
  2. AFC > 16
  3. PCOS diagnosed according to Rotterdam criteria [19, 28]: any two of the following three features: 1) oligo- or anovulation; 2) clinical and/or biochemical hyper-androgenemia; and 3) PCO-US with exclusion of other etiologies as mentioned in the NICHD criteria
  4. Previous OHSS
  5. Previous cycle cancellation due to OHSS risk
  6. Previous coasting
  7. Excessive ovarian response markers on triggering day such as high amount of middle-large follicles (> 13 follicles ≥ 11mm on triggering day) and E2 concentration (optional E2 > 14500 pmol/L on triggering day). These patients will be allocated to the high responders group.
* Untreated uterine abnormalities
* Chronic disease

C) Dual Triggering for Poor Responders

Inclusion criteria: According to Bologna criteria two of the following should be fulfilled:

* Age > 40 or other risk factor for decreased ovarian reserve (ex. ovarian surgery).
* Single abnormal test for ovarian reserve (AFC < 6 or AMH < 8 pmol/L).
* Previous poor response in previous cycle: cancellation or < 4 retrieved oocytes in response to daily 150 FSH units.

Exclusion criteria:

* Chronic disease
* Untreated uterine abnormalities
* Response consistent with normal or high responder, as defined above

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 666 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 14 days post IVF procedure
Human Chorionic Gonadotropin serum levels | 2-4 weeks post IVF procedure
Ongoing pregnancy rate | 9 months post IVF procedure
Miscarriage rate | 9 months post procedure
Ovarian hyperstimulation syndrome | 7 days post IVF procedure
  Mild OHSS:
  1. Grade 1: Abdominal distention, Ovaries <6 cm
  2. Grade 2: Abdominal distention and nausea, vomiting and diarrhea, Ovaries <6 cm
  Moderate OHSS:
  a) Grade 3: Grade II criteria and ultrasound ascites/weight gain, Ovaries 6-12 cm
  Severe OHSS:
  1. Grade 4: Ascites/hydrothorax, Ovaries >12 cm
  2. Grade 5: Ascites/hydrothorax and hypovolemia, hemoconcentration, coagulation disorder, oliguria, shock, Ovaries >12 cm
Fetal heartbeat measured by ultrasound | 2-4 weeks post IVF procedure

SECONDARY OUTCOMES:
Number of retrieved oocytes | 5 days post IVF procedure
Number of retrieved Meiosis II oocytes | 5 days post IVF procedure
Fertilization rate | 5 days post IVF procedure
Number of Day 3 embryos/eggs retrieved | 5 days post IVF procedure
Number of blastocysts/eggs retrieved | 5 days post IVF procedure

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Librach, MD, Principal Investigator — University of Toronto
Locations (1):
- Create Fertility Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tremellen K, Savulescu J. Ovarian reserve screening: a scientific and ethical analysis. Hum Reprod. 2014 Dec;29(12):2606-14. doi: 10.1093/humrep/deu265. Epub 2014 Oct 21. PMID 25336704
- [Background] Sills ES, Alper MM, Walsh AP. Ovarian reserve screening in infertility: practical applications and theoretical directions for research. Eur J Obstet Gynecol Reprod Biol. 2009 Sep;146(1):30-6. doi: 10.1016/j.ejogrb.2009.05.008. Epub 2009 May 31. PMID 19487066
- [Background] Garcia JE, Jones GS, Acosta AA, Wright G Jr. Human menopausal gonadotropin/human chorionic gonadotropin follicular maturation for oocyte aspiration: phase I, 1981. Fertil Steril. 1983 Feb;39(2):167-73. doi: 10.1016/s0015-0282(16)46814-7. PMID 6217993
- [Background] Ferraretti AP, La Marca A, Fauser BC, Tarlatzis B, Nargund G, Gianaroli L; ESHRE working group on Poor Ovarian Response Definition. ESHRE consensus on the definition of 'poor response' to ovarian stimulation for in vitro fertilization: the Bologna criteria. Hum Reprod. 2011 Jul;26(7):1616-24. doi: 10.1093/humrep/der092. Epub 2011 Apr 19. PMID 21505041
- [Background] Tarlatzis BC, Zepiridis L, Grimbizis G, Bontis J. Clinical management of low ovarian response to stimulation for IVF: a systematic review. Hum Reprod Update. 2003 Jan-Feb;9(1):61-76. doi: 10.1093/humupd/dmg007. PMID 12638782
- [Background] Lainas TG, Sfontouris IA, Papanikolaou EG, Zorzovilis JZ, Petsas GK, Lainas GT, Kolibianakis EM. Flexible GnRH antagonist versus flare-up GnRH agonist protocol in poor responders treated by IVF: a randomized controlled trial. Hum Reprod. 2008 Jun;23(6):1355-8. doi: 10.1093/humrep/den107. Epub 2008 Apr 10. PMID 18403419
- [Background] Datta AK, Eapen A, Birch H, Kurinchi-Selvan A, Lockwood G. Retrospective comparison of GnRH agonist trigger with HCG trigger in GnRH antagonist cycles in anticipated high-responders. Reprod Biomed Online. 2014 Nov;29(5):552-8. doi: 10.1016/j.rbmo.2014.08.006. Epub 2014 Aug 28. PMID 25246126
- [Background] Huber M, Hadziosmanovic N, Berglund L, Holte J. Using the ovarian sensitivity index to define poor, normal, and high response after controlled ovarian hyperstimulation in the long gonadotropin-releasing hormone-agonist protocol: suggestions for a new principle to solve an old problem. Fertil Steril. 2013 Nov;100(5):1270-6. doi: 10.1016/j.fertnstert.2013.06.049. Epub 2013 Aug 6. PMID 23931964
- [Background] Broekmans FJ, Verweij PJ, Eijkemans MJ, Mannaerts BM, Witjes H. Prognostic models for high and low ovarian responses in controlled ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2014 Aug;29(8):1688-97. doi: 10.1093/humrep/deu090. Epub 2014 Jun 5. PMID 24903202
- [Background] Klein JU, Sauer MV. Ethics in egg donation: past, present, and future. Semin Reprod Med. 2010 Jul;28(4):322-8. doi: 10.1055/s-0030-1255180. Epub 2010 Aug 3. PMID 20683796
- [Background] Prapas Y, Panagiotidis I, Kalogiannidis I, Gjata E, Papatheodorou A, Prapa S, Kasapi L, Goudakou M, Prapas N. Double GnRH-antagonist dose before HCG administration may prevent OHSS in oocyte-donor cycles: a pilot study. Reprod Biomed Online. 2010 Aug;21(2):159-65. doi: 10.1016/j.rbmo.2010.04.030. Epub 2010 Jun 2. PMID 20627811
- [Background] Melo M, Busso CE, Bellver J, Alama P, Garrido N, Meseguer M, Pellicer A, Remohi J. GnRH agonist versus recombinant HCG in an oocyte donation programme: a randomized, prospective, controlled, assessor-blind study. Reprod Biomed Online. 2009 Oct;19(4):486-92. doi: 10.1016/j.rbmo.2009.06.001. PMID 19909588
- [Background] Gonen Y, Balakier H, Powell W, Casper RF. Use of gonadotropin-releasing hormone agonist to trigger follicular maturation for in vitro fertilization. J Clin Endocrinol Metab. 1990 Oct;71(4):918-22. doi: 10.1210/jcem-71-4-918. PMID 2119392
- [Background] Humaidan P, Polyzos NP. Human chorionic gonadotropin vs. gonadotropin-releasing hormone agonist trigger in assisted reproductive technology--"the king is dead, long live the king!". Fertil Steril. 2014 Aug;102(2):339-41. doi: 10.1016/j.fertnstert.2014.04.047. Epub 2014 Jun 4. No abstract available. PMID 24907915
- [Background] Fauser BC, de Jong D, Olivennes F, Wramsby H, Tay C, Itskovitz-Eldor J, van Hooren HG. Endocrine profiles after triggering of final oocyte maturation with GnRH agonist after cotreatment with the GnRH antagonist ganirelix during ovarian hyperstimulation for in vitro fertilization. J Clin Endocrinol Metab. 2002 Feb;87(2):709-15. doi: 10.1210/jcem.87.2.8197. PMID 11836309
- [Background] Humaidan P, Bredkjaer HE, Bungum L, Bungum M, Grondahl ML, Westergaard L, Andersen CY. GnRH agonist (buserelin) or hCG for ovulation induction in GnRH antagonist IVF/ICSI cycles: a prospective randomized study. Hum Reprod. 2005 May;20(5):1213-20. doi: 10.1093/humrep/deh765. Epub 2005 Mar 10. PMID 15760966
- [Background] Kolibianakis EM, Schultze-Mosgau A, Schroer A, van Steirteghem A, Devroey P, Diedrich K, Griesinger G. A lower ongoing pregnancy rate can be expected when GnRH agonist is used for triggering final oocyte maturation instead of HCG in patients undergoing IVF with GnRH antagonists. Hum Reprod. 2005 Oct;20(10):2887-92. doi: 10.1093/humrep/dei150. Epub 2005 Jun 24. PMID 15979994
- [Background] Humaidan P, Kol S, Papanikolaou EG; Copenhagen GnRH Agonist Triggering Workshop Group. GnRH agonist for triggering of final oocyte maturation: time for a change of practice? Hum Reprod Update. 2011 Jul-Aug;17(4):510-24. doi: 10.1093/humupd/dmr008. Epub 2011 Mar 30. PMID 21450755
- [Background] Engmann L, DiLuigi A, Schmidt D, Nulsen J, Maier D, Benadiva C. The use of gonadotropin-releasing hormone (GnRH) agonist to induce oocyte maturation after cotreatment with GnRH antagonist in high-risk patients undergoing in vitro fertilization prevents the risk of ovarian hyperstimulation syndrome: a prospective randomized controlled study. Fertil Steril. 2008 Jan;89(1):84-91. doi: 10.1016/j.fertnstert.2007.02.002. Epub 2007 Apr 26. PMID 17462639
- [Background] Acevedo B, Gomez-Palomares JL, Ricciarelli E, Hernandez ER. Triggering ovulation with gonadotropin-releasing hormone agonists does not compromise embryo implantation rates. Fertil Steril. 2006 Dec;86(6):1682-7. doi: 10.1016/j.fertnstert.2006.05.049. Epub 2006 Oct 30. PMID 17074344
- [Background] Blazquez A, Guillen JJ, Colome C, Coll O, Vassena R, Vernaeve V. Empty follicle syndrome prevalence and management in oocyte donors. Hum Reprod. 2014 Oct 10;29(10):2221-7. doi: 10.1093/humrep/deu203. Epub 2014 Aug 1. PMID 25085799
- [Background] Bodri D, Guillen JJ, Trullenque M, Schwenn K, Esteve C, Coll O. Early ovarian hyperstimulation syndrome is completely prevented by gonadotropin releasing-hormone agonist triggering in high-risk oocyte donor cycles: a prospective, luteal-phase follow-up study. Fertil Steril. 2010 May 1;93(7):2418-20. doi: 10.1016/j.fertnstert.2009.08.036. Epub 2009 Oct 2. PMID 19800620
- [Background] Humaidan P, Polyzos NP, Alsbjerg B, Erb K, Mikkelsen AL, Elbaek HO, Papanikolaou EG, Andersen CY. GnRHa trigger and individualized luteal phase hCG support according to ovarian response to stimulation: two prospective randomized controlled multi-centre studies in IVF patients. Hum Reprod. 2013 Sep;28(9):2511-21. doi: 10.1093/humrep/det249. Epub 2013 Jun 9. PMID 23753114
- [Background] Griffin D, Benadiva C, Kummer N, Budinetz T, Nulsen J, Engmann L. Dual trigger of oocyte maturation with gonadotropin-releasing hormone agonist and low-dose human chorionic gonadotropin to optimize live birth rates in high responders. Fertil Steril. 2012 Jun;97(6):1316-20. doi: 10.1016/j.fertnstert.2012.03.015. Epub 2012 Apr 3. PMID 22480822
- [Background] Lin MH, Wu FS, Lee RK, Li SH, Lin SY, Hwu YM. Dual trigger with combination of gonadotropin-releasing hormone agonist and human chorionic gonadotropin significantly improves the live-birth rate for normal responders in GnRH-antagonist cycles. Fertil Steril. 2013 Nov;100(5):1296-302. doi: 10.1016/j.fertnstert.2013.07.1976. Epub 2013 Aug 28. PMID 23993928
- [Background] Griffin D, Feinn R, Engmann L, Nulsen J, Budinetz T, Benadiva C. Dual trigger with gonadotropin-releasing hormone agonist and standard dose human chorionic gonadotropin to improve oocyte maturity rates. Fertil Steril. 2014 Aug;102(2):405-9. doi: 10.1016/j.fertnstert.2014.04.028. Epub 2014 May 17. PMID 24842671
- [Background] Haas J, Zilberberg E, Dar S, Kedem A, Machtinger R, Orvieto R. Co-administration of GnRH-agonist and hCG for final oocyte maturation (double trigger) in patients with low number of oocytes retrieved per number of preovulatory follicles--a preliminary report. J Ovarian Res. 2014 Aug 2;7:77. doi: 10.1186/1757-2215-7-77. PMID 25296696
- [Background] Nastri CO, Teixeira DM, Moroni RM, Leitao VM, Martins WP. Ovarian hyperstimulation syndrome: pathophysiology, staging, prediction and prevention. Ultrasound Obstet Gynecol. 2015 Apr;45(4):377-93. doi: 10.1002/uog.14684. Epub 2015 Mar 1. PMID 25302750
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Papanikolaou EG, Humaidan P, Polyzos NP, Tarlatzis B. Identification of the high-risk patient for ovarian hyperstimulation syndrome. Semin Reprod Med. 2010 Nov;28(6):458-62. doi: 10.1055/s-0030-1265671. Epub 2010 Nov 16. PMID 21082503
- [Background] Seyhan A, Ata B, Polat M, Son WY, Yarali H, Dahan MH. Severe early ovarian hyperstimulation syndrome following GnRH agonist trigger with the addition of 1500 IU hCG. Hum Reprod. 2013 Sep;28(9):2522-8. doi: 10.1093/humrep/det124. Epub 2013 Apr 30. PMID 23633553
- [Background] Sunkara SK, Coomarasamy A, Faris R, Braude P, Khalaf Y. Long gonadotropin-releasing hormone agonist versus short agonist versus antagonist regimens in poor responders undergoing in vitro fertilization: a randomized controlled trial. Fertil Steril. 2014 Jan;101(1):147-53. doi: 10.1016/j.fertnstert.2013.09.035. Epub 2013 Nov 1. PMID 24188873
- [Background] Zivi E, Simon A, Laufer N. Ovarian hyperstimulation syndrome: definition, incidence, and classification. Semin Reprod Med. 2010 Nov;28(6):441-7. doi: 10.1055/s-0030-1265669. Epub 2010 Nov 16. PMID 21082501